CLINICAL TRIAL: NCT04697836
Title: Can Ultrasound-Guided Bilateral Cervical Plexus Block Combined With Translaryngeal Block For Tracheostomy Be An Alternative To General Anesthesia?
Brief Title: Cervical Plexus Block Combined With Translaryngeal Block for Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ayhan ŞAHİN, Asistant Prof, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Regional anesthesia
Record Dates: First submitted 2020-12-25; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Regional Anesthesia Morbidity
Keywords: Regional Anesthesia; Tracheostomy; Ultrasound

STUDY DESIGN:
Intervention Model Description: the new indication for cervical plexus block.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ST (superficial cervical plexus block combined with Translareyngeal block) (Experimental): Superficial cervical plexus block combined with Translareyngeal block Group.
  Interventions: Procedure: ST
- S (superficial cervical plexus block) (Active Comparator): Superficial cervical plexus block Group
  Interventions: Procedure: ST

INTERVENTIONS:
Procedure: ST — After a computer-generated randomization list with a 1:1 intergroup ratio, ensuring equal distribution in the two groups, 30 opaque sealed envelopes numbered 1-30 were prepared. The patients were randomly divided into the Group with bilateral CPB with 15 ml 0.5% bupivacaine or the patients with translaryngeal block with 5 ml 2% lidocaine in addition to bilateral CPB.
  Following inclusion, two research assistants, with no further involvement in the study, prepared 15mL syringes and 5 ml syringes according to the envelope's specifications. The syringes were marked with the patient's randomization number. All other investigators, staff, and patients were blinded to group allocations. Before surgery, the patients were transferred to the specified block room area monitored with 3-lead electrocardiography, pulse oximetry, and non-invasive blood pressure. All patients had two intravenous cannula lines, and then bilateral CPB block procedures were performed in awake non-sedated patients.

SUMMARY:
Current healthcare delivery models emphasize enhanced postoperative recovery (ERAS) with minimal morbidity and shorter hospital stays. Most tracheostomy cases are tumour patients. The more the patients have difficulty in breathing, the more difficult it is to anaesthetize them. Adequate intraoperative anaesthesia and postoperative analgesia with minimal sedation play an essential role in this patient model. In tracheostomy patients, moving away from the general anaesthesia option increases airway safety, and avoiding the local anaesthesia option in the incision area increases patient comfort. The purpose of this study is to assess the safety and efficacy of regional anaesthesia in tracheostomy patients.

DETAILED DESCRIPTION:
after being informed and about the study and potential risks, all patients giving written informed consent will undergo 24 hours screening period to determine the eligilibity for study entry. After a computer-generated randomization list with a 1:1 intergroup ratio, ensuring equal distribution in the two groups, 30 opaque sealed envelopes numbered 1-30 were prepared. The patients were randomly divided into the Group with bilateral CPB with 15 ml 0.5% bupivacaine or the patients with translaryngeal block with 5 ml 2% lidocaine in addition to bilateral CPB.

CPB: cervical plexus block.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-65, with American Society of Anesthesiology (ASA) classification I-III and scheduled for elective or emergency tracheostomy.
* A sufficient level of education to understand the study procedures and agree to participate in the study

Exclusion Criteria:

* inability to cooperate
* dementia,
* allergy to local anesthetics and opioids
* regular daily opioid requirements
* abuse of alcohol or medication
* local infection at the site of injection or systemic infection,
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
pain score (NRS) | 24 hours
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
pain related to incision | 24 hours
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Patient tolerance as assessed by tracheostomy cannula comfort score | 24 hours
  1. = No reaction
  2. = Slight grimacing
  3. = Heavy grimacing
  4. = Defensive movement of hands 5= Flexion of the head with defense
cough and gag score | 24 hours
  1. = None
  2. = Slight
  3. = Moderate
  4. = Severe
nausea and vomiting | 24 hours
  YES/NO
time to first analgesic demand | 24 hours from the pacu
  Time of first analgesic need within the first 24 hours 0: within the first 12 hours
  1: 12-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: AYHAN ŞAHİN, Study Director — Clinical Director
Locations (1):
- Namık Kemal University, Tekirdağ, Süleymanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Demographic and clinical features of the study groups.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: study is finished
Access Criteria: public

REFERENCES:
- [Background] Mehta AB, Syeda SN, Bajpayee L, Cooke CR, Walkey AJ, Wiener RS. Trends in Tracheostomy for Mechanically Ventilated Patients in the United States, 1993-2012. Am J Respir Crit Care Med. 2015 Aug 15;192(4):446-54. doi: 10.1164/rccm.201502-0239OC. PMID 25955332
- [Background] Bradley PJ. Treatment of the patient with upper airway obstruction caused by cancer of the larynx. Otolaryngol Head Neck Surg. 1999 May;120(5):737-41. doi: 10.1053/hn.1999.v120.a90043. PMID 10229602
- [Background] Freeman BD. Indications for and management of tracheostomy. In: Vincent JL, Abraham E, Moore FA, et al, editors. Textbook of critical care. 6th edition. Phila- delphia: Elsevier/W. B. Saunders; 2011. p. 369-72
- [Background] Moorthy SS, Gupta S, Laurent B, Weisberger EC. Management of airway in patients with laryngeal tumors. J Clin Anesth. 2005 Dec;17(8):604-9. doi: 10.1016/j.jclinane.2004.12.019. PMID 16427530
- [Background] Kim JS, Ko JS, Bang S, Kim H, Lee SY. Cervical plexus block. Korean J Anesthesiol. 2018 Aug;71(4):274-288. doi: 10.4097/kja.d.18.00143. Epub 2018 Jul 4. PMID 29969890

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT04697836/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT04697836/SAP_001.pdf